CLINICAL TRIAL: NCT00707785
Title: Effect of Vitamin A in the Treatment of Sepsis and Necrotizing Enterocolitis in Hospitalized Neonates
Brief Title: Effect of Vitamin A in the Treatment of Neonatal Sepsis and Necrotizing Enterocolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christian Coles, Assistant Professor, Department of International Health, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H.22.05.12.20.A2; 1K01DK075478-01 (NIH)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Sepsis; Necrotizing Enterocolitis; Meningitis; Pneumonia
Keywords: vitamin A; Treatment; neonates; newborn; sepsis; necrotizing enterocolitis; meningitis; pneumonia
MeSH Terms: conditions — Sepsis; Enterocolitis, Necrotizing; Meningitis; Pneumonia | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Sepsis - vitamin A
  Interventions: Dietary Supplement: Vitamin A
- 2 (Placebo Comparator): Sepsis - placebo
  Interventions: Dietary Supplement: Vitamin A
- 3 (Experimental): NEC - vitamin A
  Interventions: Dietary Supplement: Vitamin A
- 4 (Placebo Comparator): NEC - Placebo
  Interventions: Dietary Supplement: Vitamin A

INTERVENTIONS:
Dietary Supplement: Vitamin A — 50,000 IU of Vitamin A 50,000 IU of vegetable oil
  Other Names: Retinol

SUMMARY:
The purpose of the study is to determine whether vitamin A can improve survival and facilitate recovery from sepsis and necrotizing enterocolitis in hospitalized neonates.

DETAILED DESCRIPTION:
Sepsis and necrotizing enterocolitis (NEC) are leading causes of morbidity and mortality in neonates. Studies have shown that early reversal of the signs associated with severe disease is an important prognostic factor during acute illness. Vitamin A deficiency is widespread among children, including neonates, in developing countries. Vitamin A plays an important role in mediating immune responses and in maintaining epithelial integrity. For this reason vitamin A supplementation during the acute phase of neonatal infection could work synergistically with present antibiotic regimens in promoting early reversal of signs associated with adverse outcome and shorten the total duration of clinical illness. The purpose of the proposed hospital-based clinical trial is to evaluate the efficacy of vitamin A supplementation on reducing the morbidity and mortality among neonates hospitalized with sepsis (n=366) and NEC(n=150). Enrolled subjects will be randomized at the time of hospitalization to receive one dose of either 50,000 IU of vitamin A or placebo at enrollment, in addition to standard antibiotic therapy. We will compare the proportion of treatment failures in sepsis patients, the frequency of disease progression and mortality in NEC patients, and the time to clinical recovery and discharge between treatment groups. In addition, the study will determine whether vitamin A reduces pro-inflammatory cytokine levels; elevated host inflammatory cytokines are thought to contribute to the severity of both conditions. If vitamin A is found to be efficacious in the treatment of sepsis and NEC it could present a needed cost-effective approach to decreasing the global morbidity, mortality and the economic cost associated with neonatal sepsis and NEC in the developing world.

ELIGIBILITY:
Inclusion Criteria:

* newborns less than 29 days with clinical sepsis

Exclusion Criteria:

* healthy infants
* major congenital abnormalities
* known inborn error(s) of metabolism
* chronic disorders of other organs (e.g. cholestasis)
* definite or severe NEC (> stage 2)
* congenital heart disease
* Infants receiving VA supplements
* Infants requiring mechanical ventilation
* Infant is unconscious

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2006-12; Primary Completion 2011-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Disease Mortality | prospective

SECONDARY OUTCOMES:
Inflammatory cytokine concentration | prospective
Duration of inflammation | prospective
Disease progression in NEC patients | prospective

OTHER OUTCOMES:
Treatment failure | prospective
Time to recovery from severe illness | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Coles, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Dhaka Shishu Hospital, Dhaka, Bangladesh